CLINICAL TRIAL: NCT04394819
Title: The Effect of Task-oriented Electromyography-triggered Electrical Stimulation on Upper Limb Motor Function in Hemiplegic Cerebral Palsy
Brief Title: The Effect of Task-oriented EMG-triggered ES on Upper Limb Motor Function in Hemiplegic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: nihal tezel (Other Government)
Responsible Party: Sponsor-Investigator, nihal tezel, medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Organization: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Other Study IDs: DiskapiYBERHPTR
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy, Spastic
Keywords: cerebral palsy; task-oriented training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- experimental and control groups: Task-oriented EMG-triggered ES treatment will be applied to the experimental group 2 days a week for 5 weeks and will continue with conventional physiotherapy.
  The control group will only continue conventional physiotherapy treatment.
  Interventions: Other: electromyography-triggered electrical stimulation

INTERVENTIONS:
Other: electromyography-triggered electrical stimulation — All treatments were planned as 2 sessions per week, for a total of 10 sessions for 5 weeks. For EMG-trigger-ES application, dual-channel Nu-Tek® brand, Maxi plus 2 Model EMG-trigger-BF-ES Device in our clinic was planned to be used. With EMG-triggered-ES application, while the patient is in a sitting position, shoulder adduction, and the elbow is 90 degrees of flexion and pronation, the patient will extend to the ball of 5 cm in diameter, which is placed as far as the distance between the acromion and the 3rd toe, and then the finger-wrist active extension will be stimulated and then It was planned to apply the ball to be grasped. One of the two 5x5 cm superficial square electrodes of the device was planned to be placed on the extensor carpi radialis and extensor digitorum Communis and the other 2 cm distal.

SUMMARY:
The purpose of our study; to investigate the effects of EMG-induced ES treatment on hand functions, muscle strength, and quality of life in patients with hemiplegic CP.

DETAILED DESCRIPTION:
Upper limb spasticity greatly affects the hand functions of patients with cerebral palsy (CP) and impairs quality of life. The most important goal in rehabilitation; despite the existing deficiencies, the highest level of functional independence of the patient is to increase the quality of life. EMG-triggered biofeedback electrical stimulation (EMG-triggered-BF-ES) increases the patient's active participation and motivation in rehabilitation, creates visual or auditory BF, provides muscle reeducation, decreases spasticity, prevents atrophies and increases joint mobility and increases muscle functionality by increasing the patient's functionality. There are areas of use the EMG-triggered-BF-ES such as cerebrovascular disease (CVO), spinal cord injury, and CP. When the literature is examined; studies were found to be few, and no study evaluating the upper extremity was found in children with CP. The purpose of our study is the investigation of the effects of EMG-triggered-BF-ES treatment applied on hand functions, muscle strength, and quality of life in patients with CP.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of CP
* age between 4 and 18 year
* at least 10° of the active wrist and finger extension in the affected limb but less than normal
* upper limb spasticity (shoulder, elbow, wrist, and fingers) less than or equal to grade 2 according to the modified Ashworth scale (MAS)
* should be able to receive command

Exclusion Criteria:

* Mental retardation
* Passive range of motion (ROM) limitation in the upper extremity
* Sensory impairment in the upper extremity
* The visual and auditory deficit in the upper extremity
* MAS is more than 3.
* Botulinum toxin application to the upper limb in the last 6 months
* Any surgical application to the upper limb in the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — age between 4-18
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The Cerebral Palsy Quality of Life Questionnaire (CPQoL) | within 3 months
  Health condition-specific questionnaire designed for measuring QOL in children with cerebral palsy (CP). It consists of a caregiver and a child survey. It is used for the evaluation of Sp cases between the ages of 4-12.
Action Research Arm Test (ARAT) | within 3 months
  The ARAT consists of four subscales: grasp, grip, pinch, and gross movement. It contains 19 tasks, and each task is scored on a four-point scale (0, can perform no part of the test; 1, performs test partially; 2, completes test but takes abnormally long time or has great difficulty; and 3, performs test normally).

SECONDARY OUTCOMES:
nine hole peg test (9-HPT) | at the beginning, at the 5th week, and at the 3rd-month visit.
  9-HPT test is a standardized,quantitative assesment used to measure finger dexterity.
hydraulic hand dynamometer | at the beginning, at the 5th week, and at the 3rd-month visit.
  Patients were encouraged to press as firmly as possible. Three consecutive measurements were performed. The average of the measurements was recorded in kilogram (kg).

CONTACTS AND LOCATIONS:
Locations (1):
- DiskapiYBERH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Electromyography-Triggered Electrical Muscle Stimulation for Children with Cerebral Palsy: A Pilot Study — https://journals.lww.com/pedpt/Abstract/1991/00340/Electromyography_Triggered_Electrical_Muscle.4.aspx
- See also: Electrical stimulation in cerebral palsy: a review of effects on strength and motor function — https://pubmed.ncbi.nlm.nih.gov/14995090
- See also: Therapeutic effects of functional electrical stimulation of the upper limb of eight children with cerebral palsy — https://www.ncbi.nlm.nih.gov/pubmed/11104342
- See also: Therapeutic functional electrical stimulation in hemiplegic cerebral palsy — https://pubmed.ncbi.nlm.nih.gov/24185362